CLINICAL TRIAL: NCT04869176
Title: Effect of Caffeine for Apnoea Treatment on Heart Rate Variability in Newborns
Brief Title: Effect of Caffeine on Heart Rate Variability in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Petja Fister, Assist. Prof. Petja Fister, MD, PhD, University of Ljubljana
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0120-458/2016-3
Record Dates: First submitted 2021-03-20; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Caffeine; Heart Rate Variability; Apnoea of Newborn; Newborn
Keywords: newborn; heart rate variability; caffeine; bed tilt; autonomic nervous system
MeSH Terms: interventions — Electrocardiography; Electrocardiography, Ambulatory; caffeine citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On Caffeine, maintenance dose (Experimental): During receiving maintenance dose of 5 mg/kg caffeine citrate (i.e. 2,5 mg/kg caffeine) in the form of solution, orally or intravenously, Holter electrocardiogram and vital functions were monitored for 40 minutes.
  Interventions: Diagnostic Test: Electrocardiogram; Diagnostic Test: Monitoring of vital functions; Drug: Caffeine Citrate 5 mg/kg
- Off caffeine (Experimental): 100 hours after caffeine withdrawal Holter electrocardiogram and vital functions were monitored for 40 minutes.
  Interventions: Diagnostic Test: Electrocardiogram; Diagnostic Test: Monitoring of vital functions

INTERVENTIONS:
Diagnostic Test: Electrocardiogram — Recording of the electrical activity of the heart during sleep; sleep phases were evaluated. The bed was initially in horizontal position and tilted for 30° head-up after 20 minutes of continuous tracing.
  Other Names: Holter ECG
Diagnostic Test: Monitoring of vital functions — Measuring of heart rate, breathing frequency, arterial oxygen saturation and body temperature while recording ECG.
Drug: Caffeine Citrate 5 mg/kg — Caffeine in the form of suspension was given to the newborns.
  Arms: On Caffeine, maintenance dose

SUMMARY:
The aim of this study was to evaluate the impact of caffeine treatment, given either orally or intravenously, on heart rate variability in newborns. In addition, the investigators sought for a potential association between caffeine treatment and vital functions.

DETAILED DESCRIPTION:
At Neonatal Department of University Medical Centre Ljubljana caffeine is used to treat neonatal apnoea. It has known affects on central nervous and cardiovascular systems, but little is known about the impact of caffeine intake on heart rate variability (HRV) in newborns.

In this study, the investigators performed measurements on one sample of 25 newborns with apnoea who had been admitted to the Neonatal Department of University Medical Centre Ljubljana and treated with caffeine citrate. The treatment regimen consisted of caffeine citrate of a loading dose of 20 mg/kg of body mass, followed by a daily maintenance dose of 5 mg/kg after 24 hours. The investigators measured parameters of HRV in two situations: while the treatment with caffeine citrate was ongoing and after the treatment was withdrawn. The newborns served as controls. Electrical activity of the heart was measured with a Holter ECG while the newborn was sleeping in supine position, first without a bed tilt and afterwards with a 30° head-up tilt. Simultaneously was evaluated the alertness of the newborn and measured their physiological variables (the breathing frequency, the heart rate, the arterial oxygen saturation, and the body temperature).

All parents were given their written consent for their child to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* newborns with apnoea treated with caffeine citrate
* newborns whose parents have signed the informed consent form

Exclusion Criteria:

* severe perinatal hypoxia
* infection
* liver or renal insufficiency
* neurological disorders
* congenital anomalies

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Association between caffeine treatment and total power (TP) spectrum of HRV | During Procedure
  While the newborn was sleeping, the electrical activity of the heart was recorded by using ECG Holter. TP (ms2) was obtained from a suitable 5-minute ECG segment analysed by fast Fourier transform, using the Vision Premier Programme for each bed tilt. The values were compared across the two arms of the study, using student's t-test for comparisons of normally distributed variables, and Wilcoxon signed-rank test for abnormally distributed data.
Association between caffeine treatment and high frequency (HF) spectrum of HRV | During Procedure
  While the newborn was sleeping, the electrical activity of the heart was recorded by using ECG Holter. HF (ms2) was obtained from a suitable 5-minute ECG segment analysed by fast Fourier transform, using the Vision Premier Programme for each bed tilt. The values were compared across the two arms of the study, using student's t-test for comparisons of normally distributed variables, and Wilcoxon signed-rank test for abnormally distributed data.
Association between caffeine treatment and low frequency (LF) spectrum of HRV | During Procedure
  While the newborn was sleeping, the electrical activity of the heart was recorded by using ECG Holter. LF (ms2) was obtained from a suitable 5-minute ECG segment analysed by fast Fourier transform, using the Vision Premier Programme for each bed tilt. The values were compared across the two arms of the study, using student's t-test for comparisons of normally distributed variables, and Wilcoxon signed-rank test for abnormally distributed data.

SECONDARY OUTCOMES:
The correlation between postmenstrual age and total power (TP) spectrum of HRV | During Procedure
  While the newborn was sleeping, the electrical activity of the heart was recorded by using ECG Holter. TP (ms2) was obtained from a suitable 5-minute ECG segment analysed by fast Fourier transform, using the Vision Premier Programme for each bed tilt. The correlation between HRV parameters and postmenstrual age was tested with the Pearson correlation coefficient.
The correlation between postmenstrual age and high frequency (HF) spectrum of HRV | During Procedure
  While the newborn was sleeping, the electrical activity of the heart was recorded by using ECG Holter. HF (ms2) was obtained from a suitable 5-minute ECG segment analysed by fast Fourier transform, using the Vision Premier Programme for each bed tilt. The correlation between HRV parameters and postmenstrual age was tested with the Pearson correlation coefficient.
The correlation between postmenstrual age and low frequency (LF) spectrum of HRV | During Procedure
  While the newborn was sleeping, the electrical activity of the heart was recorded by using ECG Holter. LF (ms2) was obtained from a suitable 5-minute ECG segment analysed by fast Fourier transform, using the Vision Premier Programme for each bed tilt. The correlation between HRV parameters and postmenstrual age was tested with the Pearson correlation coefficient.
The effect of caffeine on heart rate | During Procedure
  Heart rate (beats per minute) was obtained from the segments, recorded by ECG Holter and analysed by the Vision Premier Programme. The selected segments corresponded to the segments HRV parameters were obtained for each bed tilt. The values were compared across the two arms of the study.
The effect of caffeine on breathing frequency | During Procedure
  Breathing frequency (breaths per minute) was determined manually by observing the chest movement. The measurement was performed three times while the newborn was sleeping for each bed tilt. The values were compared across the two arms of the study.
The effect of caffeine on arterial oxygen saturation | During Procedure
  Arterial oxygen saturation (percent) was performed by a pulse oximeter attached to the right hand. The arterial oxygen saturation value was noted three times with the corresponding breathing frequency while the newborn was sleeping for each bed tilt. The values were compared across the two arms of the study.
The effect of caffeine on body temperature | During Procedure
  Body temperature (degree Celsius) was measured by a frontal non-contact infrared thermometer three times for each bed tilt while the newborn was sleeping. The values were compared across the two arms of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Petja Fister, MD, PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/76/NCT04869176/Prot_SAP_000.pdf